CLINICAL TRIAL: NCT06885307
Title: Construction of a Multi-center Clinical Research Collaboration Network for Children with Congenital Heart Disease in China
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kun Sun, Professor of Department of Pediatric Cardiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2024-159-1
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Congenital Heart Disease (CHD); Database
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project intends to unite the representatives of typical congenital heart disease hospitals in various provinces and cities across the country to jointly establish a multi-center clinical research collaboration network for children with congenital heart disease in China, establish a platform and mechanism for the collection and sharing of data on children with congenital heart disease in China, and create a real-world public database of children with congenital heart disease in China that benchmarks the international level, so as to provide a solid data foundation for high-quality research on children with congenital heart disease in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-18 years, regardless of gender;
2. Patients diagnosed with congenital heart disease confirmed by cardiac ultrasound examination;

Exclusion Criteria:

None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with congenital heart disease confirmed by cardiac ultrasound examination
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of condition | Extract the discharge prognosis in the discharge summary after the hospitalization at the time of surgery
  The discharge records were extracted and written by the attending doctor, and the values were divided into cured, improved, unhealed, and died

CONTACTS AND LOCATIONS:
Overall Officials: Kun Sun, MD, Principal Investigator — Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai, 200092, China
Locations (6):
- China (6):
  - Wuhan Children's Hospital (Wuhan Maternal and Child Healthcare Hospital), Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qinghai Women & Children'S Hospital, Xining, Qinghai
  - Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Kunming Children's Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan